CLINICAL TRIAL: NCT05065658
Title: Posaconazole for the Prevention of COVID-19 Associated Pulmonary Aspergillosis in Critically-Ill Patients: A European Multicenter Case-Control Study
Brief Title: Posaconazole Prophylaxis for CAPA Prevention in Critically-Ill Patients
Acronym: POSACOVID
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 32-296 ex 19/20
Record Dates: First submitted 2021-09-09; First posted 2021-10-04 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: COVID-19 Respiratory Infection; Aspergillosis
MeSH Terms: conditions — Aspergillosis | interventions — posaconazole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Critically-ill COVID-19 patients receiving posaconazole prophylaxis
  Interventions: Drug: Posaconazole
- Critically-ill COVID-19 patients without antifungal prophylaxis

INTERVENTIONS:
Drug: Posaconazole — Intravenous posaconazole prophylaxis
  Groups: Critically-ill COVID-19 patients receiving posaconazole prophylaxis

SUMMARY:
COVID-19 associated pulmonary aspergillosis (CAPA) is considered a potentially life-threatening infection in critically ill COVID (Corona Virus disease)-19 patients. This study will investigate the efficacy of mold-active prophylaxis with posaconazole for patients with severe SARS (severe acute respiratory syndrome)-CoV-2 infection admitted to the ICU (intensive care unit) in a multi-center case-control study in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years)
* PCR (polymerase chain reaction) -confirmed SARS-CoV-2 infections based on nasopharyngeal swab (NPS), oropharyngeal swab (OPS), tracheal aspirate (TA), bronchial aspirate (BA), or bronchoalveolar lavage fluid (BALF) within 14 days prior to ICU admission or within 72 hours following ICU admission due to severe COVID-19 infection
* Radiographic imaging consistent with SARS-CoV-2 infection (e.g. atypical pneumonia, organizing pneumonia, ground glass opacities) or ARDS within 7 days of diagnosis of SARS-CoV-2 infection

Exclusion Criteria:

* Patients with a diagnosis of invasive aspergillosis/detection of Aspergillus spp. by culture from sputum, TA, BA, or BALF or positive GM from serum, TA, or BALF at baseline (=ICU admission)
* History of invasive aspergillosis within the prior six months
* Patients that are being treated with mold-active antifungal agents for invasive aspergillosis or another invasive fungal infection
* Patients that are being treated with mold-active antifungal agents for invasive aspergillosis or another invasive fungal infection
* Death or transfer to general ward within 48 hours of ICU admission
* Antifungal prophylaxis other than posaconazole (e.g. inhaled amphotericin B)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of patients admitted to the ICU because of severe SARS-CoV-2 infections, who are requiring mechanical ventilation and receive dexamethasone as part of their COVID-19 ARDS treatment in medical centers in i) Graz, Austria (cases), and ii) Genoa, Italy, and iii) Rennes, France (all controls).
  Posaconazole prophylaxis for ICU patients with severe COVID-19 requiring ICU admission due to ARDS has been introduced in Graz in July 2020, and cases from Graz will be matched with controls from Rennes and Genoa (matching for days on mechanical ventilation at baseline, Apache II score, age, dexamethasone dosage, and underlying disease).
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Medical University of Graz, Graz, Styria, Austria
- University of Rennes, Rennes, France
- San Martino Polyclinic Hospital IRCCS, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Prattes J, Giacobbe DR, Marelli C, Signori A, Dettori S, Cattardico G, Hatzl S, Reisinger AC, Eller P, Krause R, Reizine F, Bassetti M, Gangneux JP, Hoenigl M. Posaconazole for Prevention of COVID-19-Associated Pulmonary Aspergillosis in Mechanically Ventilated Patients: A European Multicentre Case-Control Study (POSACOVID). Mycoses. 2025 Jan;68(1):e70023. doi: 10.1111/myc.70023. PMID 39800852

RESULTS

PARTICIPANT FLOW:
Groups:
- COVID-19 Patients With Acute Respiratory Failure Receiving Posaconazole Prophylaxis (Center 1): Cases: Intravenous posaconazole prophylaxis
- COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 2); COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 3): Controls: Standard of care (no antifungal prophylaxis)
Period: Overall Study
Arm/Group | COVID-19 Patients With Acute Respiratory Failure Receiving Posaconazole Prophylaxis (Center 1) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 2) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 3)
Started | 83 | 83 | 83
Completed | 83 | 83 | 83
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- COVID-19 Patients With Acute Respiratory Failure Receiving Posaconazole Prophylaxis (Center 1): Cases: Subjects with COVID-19 associated ARF who received intravenous posaconazole prophylaxis upon ICU admission in addition to standard of care treatment
- COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 2); COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 3): Controls: Subjects with COVID-19 associated ARF who did not receive antifungal prophylaxis in addition to standard of care treatment
- Total: Total of all reporting groups
Arm/Group | COVID-19 Patients With Acute Respiratory Failure Receiving Posaconazole Prophylaxis (Center 1) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 2) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 3) | Total
Number analyzed (Participants) | 83 | 83 | 83 | 249
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [58 to 71] | 65 [57 to 72] | 66 [61 to 71] | 65 [58 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 54 | 165
  Male | 27 | 28 | 29 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race data were not collected Population: Race data were not collected
Region of Enrollment [Number; unit: participants]
  Austria | 83 | 0 | 0 | 83
  Italy | 0 | 83 | 0 | 83
  France | 0 | 0 | 83 | 83
Tocilizumab Treatment [Count of Participants; unit: Participants] | 2 | 3 | 1 | 6
Systemic glucocorticoid treatment [Count of Participants; unit: Participants] | 83 | 83 | 83 | 249

OUTCOME MEASURES:

1. Primary Outcome: Incidence of COVID-19 Associated Pulmonary Aspergillosis (CAPA)
Description: Compare the incidence of CAPA at time of discharge from the ICU in those who received posaconazole compared to controls who did not
Time Frame: ICU admission to ICU discharge. On average 20 days
Measure: Number; unit: Cases per 1000 ICU days
Arm/Group | COVID-19 Patients With Acute Respiratory Failure Receiving Posaconazole Prophylaxis (Center 1) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 2) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 3)
Number analyzed (Participants) | 83 | 83 | 83
Cases per 1000 ICU days | 1.69 | 0.84 | 7.18

2. Secondary Outcome: Risk Factors for CAPA Development (EORTC/MSGERC)
Description: This Outcome Measure examines whether the presence of an EORTC/MSGERC-defined risk factor at ICU admission is associated with an increased risk of developing COVID-19-associated pulmonary aspergillosis (CAPA) during the ICU stay. The analysis is conducted using a cohort of patients admitted to the ICU, tracking the development of CAPA from ICU admission to ICU discharge.
  For this purpose, the number of subjects who had underlying EORTC/MSGERC risk factors present at ICU admission was collected and used as a parameter in a multivariate logistic model to assess the association with an increased risk for CAPA development.
Time Frame: ICU admission to ICU discharge. On average 20 days
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Patients With Acute Respiratory Failure Receiving Posaconazole Prophylaxis (Center 1) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 2) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 3)
Number analyzed (Participants) | 83 | 83 | 82
Participants | 8 | 7 | 4

3. Secondary Outcome: Risk Factors for CAPA Development (ECMO)
Description: This Outcome Measure examines whether the need for extracorporal membrange oxygenation (ECMO) treatment during ICU admission is associated with an increased risk of developing COVID-19-associated pulmonary aspergillosis (CAPA) during the ICU stay. The analysis is conducted using a cohort of patients admitted to the ICU, tracking the development of CAPA from ICU admission to ICU discharge.
  For this purpose, the number of subjects who required ECMO treatment during ICU stay was collected and used as a parameter in a multivariate logistic model to assess the association with an increased risk for CAPA development.
Time Frame: ICU admission to ICU discharge. On average 20 days
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Patients With Acute Respiratory Failure Receiving Posaconazole Prophylaxis (Center 1) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 2) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 3)
Number analyzed (Participants) | 83 | 83 | 83
Participants | 13 | 2 | 4

ADVERSE EVENTS:
Time Frame: From ICU admission to Day 90
Arm/Group | COVID-19 Patients With Acute Respiratory Failure Receiving Posaconazole Prophylaxis (Center 1) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 2) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 3)
All-Cause Mortality (participants affected / at risk) | 60/83 | 14/83 | 38/83
Serious Adverse Events (participants affected / at risk) | 83/83 | 83/83 | 83/83
Other Adverse Events (participants affected / at risk) | 0/83 | 0/83 | 0/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVID-19 Patients With Acute Respiratory Failure Receiving Posaconazole Prophylaxis (Center 1) (N=83) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 2) (N=83) | COVID-19 Patients With Acute Respiratory Failure Without Antifungal Prophylaxis (Center 3) (N=83)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 83 (83) | 83 (83) | 83 (83)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT05065658/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT05065658/SAP_001.pdf